CLINICAL TRIAL: NCT04958304
Title: Moderna mRNA-1273 Observational Pregnancy Outcome Study
Brief Title: Moderna COVID-19 Vaccine mRNA-1273 Observational Pregnancy Outcome Study
Status: Terminated | Type: Observational
Why Stopped: Study has been terminated and replaced due to low enrollment.
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: mRNA-1273-P902
Record Dates: First submitted 2021-07-09; First posted 2021-07-12 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: SARS-CoV-2
Keywords: mRNA-1273; mRNA-1273 vaccine; SARS-CoV-2; SARS-CoV-2 Vaccine; Coronavirus; Virus Diseases; Messenger RNA; COVID-19; COVID-19 Vaccine; Moderna
MeSH Terms: conditions — Coronavirus Infections; Virus Diseases; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 21 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Moderna COVID-19 Vaccine in Pregnant Women: The Moderna COVID-19 Vaccine Pregnancy Registry will collect primary data from pregnant women who have received the Moderna COVID-19 vaccine and their healthcare providers (HCPs).

SUMMARY:
The main goal of this study is to evaluate the outcomes of pregnancy in females exposed to the Moderna COVID-19 vaccine (mRNA-1273) during pregnancy.

DETAILED DESCRIPTION:
The Moderna COVID-19 Vaccine Pregnancy Registry will collect and analyze information on the potential impact of exposure to the Moderna COVID-19 vaccine on pregnancy and birth outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Currently pregnant
* The outcome of pregnancy (that is, pregnancy loss or live birth) must not be known at entry.
* Agrees to electronically sign the release of medical information form permitting the study to contact her HCPs (for example, primary care provider [PCP], obstetrician, nurse midwife) and the infant's HCP (for example, pediatrician) for medical information.
* Received the Moderna COVID-19 vaccine at any point from 28 days prior to last menstrual period (LMP) throughout pregnancy.

Exclusion Criteria:

* Participant has received any other COVID-19 vaccines at any point from 28 days prior to LMP throughout pregnancy.
* Women currently participating in another investigational device or drug study, currently taking an investigational medicinal product, or having taken an investigational product within 28 days prior to LMP or during pregnancy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women who have been exposed the Moderna COVID-19 vaccine during the 28 days prior to their LMP or at any time during pregnancy are eligible for this exposed cohort.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-09-22 (Actual); Study Completion 2023-09-22 (Actual)

PRIMARY OUTCOMES:
Number of Participants Having Infants With Suspected Major and Minor Congenital Malformations | Up to 1 year of infant age
  Major malformations are those that have significant medical, social or cosmetic consequences, and typically require surgical intervention or are life-threatening (for example, cleft lip, spina bifida).
Number of Participants With Any Pregnancy Complications | From end of first trimester (approximately 14 weeks) up to mid-third trimester (approximately 34 weeks)
  Pregnancy complications may include preeclampsia, eclampsia, pregnancy-induced hypertension, antenatal bleeding, preterm labor, gestational diabetes, dysfunctional labor, premature rupture of membranes, placenta previa, postpartum hemorrhage, small-for-gestational-age (SGA) fetus and intrauterine growth restriction (IUGR), and non-reassuring fetal status.
Number of Participants With Any Pregnancy Outcomes | Approximately 4 weeks after expected date of delivery (EDD)
  Pregnancy outcomes may include spontaneous abortions, fetal death or stillbirth, live birth, elective or therapeutic pregnancy terminations, preterm birth, ectopic pregnancies, molar pregnancies, maternal death, and COVID-19 diagnosis.
Number of Participants With Infant Outcomes | Up to 1 year of infant age
  Infant outcomes may include minor congenital malformations, size of gestational age, low birth weight, size for age, failure to thrive, hospitalization of infants, neonatal death, perinatal death, neonatal encephalopathy, respiratory distress in the newborn, neonatal/infant infection, infant death, and infant developmental milestones.

CONTACTS AND LOCATIONS:
Locations (1):
- IQVIA Call Center for United States and Canada, Durham, North Carolina, United States